CLINICAL TRIAL: NCT00835549
Title: A Relative Bioavailability Study of Cefdinir for Oral Suspension 250 mg/5mL Under Non-Fasting Conditions
Brief Title: Cefdinir for Oral Suspension 250 mg/5mL, Non-fasting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B056502
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Cefdinir; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Cefdinir for oral suspension 250 mg/5mL
- 2 (Active Comparator)
  Interventions: Drug: OMNICEF® for oral suspension 250 mg/5mL

INTERVENTIONS:
Drug: Cefdinir for oral suspension 250 mg/5mL — 1 x 250 mg/5mL, single-dose non-fasting
  Arms: 1
Drug: OMNICEF® for oral suspension 250 mg/5mL — 1 x 250 mg/5mL, single-dose non-fasting
  Arms: 2

SUMMARY:
The objective of this study is to compare the relative bioavailability of cefdinir for oral suspension 250 mg/5mL (manufactured and distributed by TEVA Pharmaceuticals USA) with that of OMNICEF® for oral suspension, 250 mg/5mL (Abbott) in healthy, adult, non-smoking subjects under non-fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* All subjects selected for this study will be non-smokers at least 18 years of age. Subjects will have a BMI (body mass index) between 19 kg/m² and 30 kg/m² (inclusive).
* Each subject will be given a general physical examination within 28 days of initiation of the study. Such examination includes but is not limited to blood pressure, general observations, and history.
* Each female subject will be given a serum pregnancy test as part of the pre-study screening process.
* Adequate blood and urine samples should be obtained within 28 days before beginning of the first period and at the end of the trial for clinical laboratory measurements.

Clinical laboratory measurements will include the following:

* Hematology: hemoglobin, hematocrit, red blood cell count, platelets, and white blood cell count (with differential).
* Clinical Chemistry: creatinine, BUN, glucose, SGOT, SGPT, bilirubin, and alkaline phosphatase.
* Urine Analysis: pH, specific gravity, protein, glucose, ketones, bilirubin, occult blood, and cells.
* HIV Screen
* Hepatitis-B, C Screen
* Drugs of Abuse Screen: pre-study and at each dosing period check-in

Subjects will be selected if all above are normal. Electrocardiograms of all participating subjects will be recorded before initiation of the study and filed with each subject's case report forms.

Exclusion Criteria:

* Subjects with a history of alcoholism or drug addiction (during past 2 years) or serious gastrointestinal, renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma (during past 5 years), diabetes, psychosis or glaucoma will not be eligible for this study.
* Subjects whose clinical laboratory test values are outside the reference range may be retested at the discretion of the clinical investigator. If the clinical values are outside the range on retesting, the subject will not be eligible to participate in the study unless the clinical investigator deems the result to not be significant.
* Subjects who have a history of allergic responses to the class of drug being tested (including penicillin, any penicillin derivative, or any cephalosporin product) should be excluded from the study.
* All subjects will have urine/saliva samples assayed for the presence of drugs of abuse as part of the clinical laboratory screening procedures and at each study period check-in. Subjects found to have urin/saliva concentrations of any of the tested drugs will not be allowed to participate.
* Subjects should not have donated blood and/or plasma for at least thirty (30) days prior to the first dosing of the study.
* Subjects who have taken any investigational drug within thirty (30) days prior to the first dosing of the study will not be allowed to participate.
* Female subjects who are pregnant, breast-feeding, or who are likely to become pregnant during the study will not be allowed to participate. Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable barrier method (e.g. condom, IUD) of contraception during the course of the study (first dosing until last blood collection) or they will not be allowed to participate. Subjects who have used implanted or injected hormonal contraceptives anytime during the 6 months prior to study dosing, or used oral hormonal contraceptives within 14 days before dosing will not be allowed to participate.
* All female subjects will be screened for pregnancy at check-in each study period. Subjects with positive or inconclusive results will be withdrawn from the study.
* Subjects who do not tolerate venipuncture will not be allowed to participate.
* Subjects who use tobacco in any form will not be eligible to participate in the study. Three months abstinence is require.

Subjects who have difficulty fasting or consuming the standard meals will not be allowed to participate.

* Subjects who have had a clinically significant illness within 4 weeks prior to the first dosing of the study will not be allowed to participate.

Subjects who have used a known hepatic enzyme inducer or inhibitor within 30 days prior to the first dosing of the study will not be allowed to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-03; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soran Hong, M.D., Principal Investigator — Novum Pharmaceutical Research Services
Locations (2):
- United States (2):
  - Novum Pharmaceutical Research Services, Houston, Texas
  - Bioassay Laboratory, Inc., Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Cefdinir (Test) First: 250mg/5mL Cefdinir for Oral Suspension test product dosed in first period followed by 250mg/5mL Omnicef® for Oral Suspension reference product dosed in the second period.
- Omnicef® (Reference) First: 250mg/5mL Omnicef® for Oral Suspension reference product dosed in first period followed by 250mg/5mL Cefdinir for Oral Suspension test product dosed in the second period.
Period: First Intervention
Arm/Group | Cefdinir (Test) First | Omnicef® (Reference) First
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Washout of 7 Days
Arm/Group | Cefdinir (Test) First | Omnicef® (Reference) First
Started | 16 | 16
Completed | 14 | 16
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Second Intervention
Arm/Group | Cefdinir (Test) First | Omnicef® (Reference) First
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cefdinir (Test) First | Omnicef® (Reference) First | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 11 | 9 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 11 | 10 | 21
  White | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 13 | 10 | 23
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration)
Description: Bioequivalence based on Cmax.
Time Frame: Blood samples collected over a 14 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cefdinir (Test): 250mg/5mL Cefdinir for Oral Suspension test product dosed in either period.
- Omnicef® (Reference): 250mg/5mL Omnicef® for Oral Suspension reference product dosed in either period.
Arm/Group | Cefdinir (Test) | Omnicef® (Reference)
Number analyzed (Participants) | 30 | 30
ng/mL | 1477.573 (573.068) | 1484.677 (531.404)
Statistical Analysis 1: Comparison: Cefdinir (Test) vs Omnicef® (Reference); Test type: Non-Inferiority or Equivalence — The ANOVA model containing factors for sequence of products, subjects within sequence, periods, and products was utilized in comparing the effects between the test and reference products. Differences were declared statistically significant at the 5% level (p<0.05); Ratio of the T/R geometric mean x 100 = 98.6, 90% CI [94.8 to 102] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference and test product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on AUC0-t.
Time Frame: Blood samples collected over a 14 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cefdinir (Test) | Omnicef® (Reference)
Number analyzed (Participants) | 30 | 30
ng*h/mL | 8009.082 (3066.97) | 7851.736 (2911.323)
Statistical Analysis 1: Comparison: Cefdinir (Test) vs Omnicef® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 102, 90% CI [98.5 to 105] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on AUC0-inf.
Time Frame: Blood samples collected over a 14 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cefdinir (Test) | Omnicef® (Reference)
Number analyzed (Participants) | 30 | 30
ng*h/mL | 8103.237 (3123.887) | 7933.332 (2957.041)
Statistical Analysis 1: Comparison: Cefdinir (Test) vs Omnicef® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 102, 90% CI [98.7 to 105] — [estimate comment as in outcome 1, analysis 1]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.